CLINICAL TRIAL: NCT02764463
Title: Clinical Survival of Indirect, Lateral-posterior 3-unit Occlusal-retained Fiber-reinforced Composite Fixed Dental Prosthesis: 15-years Follow-up
Brief Title: 15 Years Control of Fiber Reenforced Composite Fixed Partial Dentures
Acronym: FRCPDs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: BNM Clinic and Research (Other)
Responsible Party: Principal Investigator, Nicola Barabanti, DMD, BNM Clinic and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRCPDS15Y
Record Dates: First submitted 2016-03-15; First posted 2016-05-06 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Prosthodontics E06.780
Keywords: Fiber Reinforced Composites; Resin cements; Survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FRCFPDs (Other): Fiber reenforced Composite Fixed Partial Dentures
  Interventions: Device: Fiber Reinforced Composite Fixed Partial Dentures

INTERVENTIONS:
Device: Fiber Reinforced Composite Fixed Partial Dentures — All restorations were made indirectly on a plaster model using unidirectional E-glass fibers (Vectris- Ivoclar Vivadent, , liechtenstein) in combination with a laboratory resin composite (Signum, Heraeus-Kulzer)
  Other Names: FRCPDs

SUMMARY:
This prospective clinical study evaluated the performance of indirect, posterior occlusal-retained, fiber-reinforced-composite restorations.

Methods: Between June 1999 and June 2000, a total of 58 patients aged between 33 and 62 years old ( 33 male, 25 female) received 65 FCRFPD prosthesis.

All restorations were made indirectly on a plaster model using unidirectional E-glass fibers (Vectris- Ivoclar Vivadent, liechtenstein) in combination with a laboratory resin composite (Signum, Heraeus-Kulzer) and cemented according to the instructions of resin cement Variolink II (Ivoclar Vivadent). After baseline recordings, patients were followed at 6 months and thereafter annually up to 15 years. The evaluation protocol involved technical (chipping, debonding or fracture of tooth/restoration) and biological failures (caries).

DETAILED DESCRIPTION:
As of January 1999, FRC FDPs are offered as alternative to other conventional therapy options at the Department where the study was conducted. Between June-1999 and June-2000, 58 patients aged between 33 and 62 years old (25 females, 33 males, mean age: 47) received 65 indirect posterior FRC FDPs. Before enrolment in the trial, all patients were provided with a written informed consent Information was given to each patient regarding the alternative treatment options. The inclusion criteria were as follows: all subjects were required to be at least 18 years old, able to read and sign the informed consent document, physically and psychologically able to tolerate conventional restorative procedures, having no active periodontal or pulpal diseases, having no primary caries, not allergic to resin-based materials, not pregnant or nursing, having antagonist teeth opposing the FRC FDP to be restored, willing to return for follow-up examinations as outlined by the investigators. The patients who had more absent teeth than the tooth to be replaced in the rest of the dentition or those having diastemas were not excluded.

All the restorations were performed by a single operator, selected considering his clinical experience (>10 years since graduation).

All FDPs replaced one missing tooth and bonded to two adjacent abutment teeth were used for retention. No cantilever FDPs were involved.

Treatment was performed in two sessions: 1) Teeth preparation and Impression taking and model analysis, 2) Try-in, cementation and polishing of the FDP.

In the first session, after an accurate evaluation of spaces and residual dental tissues and the acceptance of this type of treatment by the patient, pillar teeth were prepared using diamond bur on high speed handpiece with mesio-occlusal, disto-occlusal, MOD, onlay or overlay preparations according to each clinical situation. Cavity preparation is required not only to remove all carious tissue, but to create a minimal space necessary to the glass fibers to support occlusal loads. According to "Munack" a cavity with 2x2mm occlusal surface and 2mm depth is able to support a 600N masticatory stress before breaking, and by increasing depth to 4mm we can reach 700N.

All cavity designs are realized following these criteria:

minimum preparation depth of 2.5mm minimum cavity width of 2mm divergent proximal boxes bucco-lingual width of proximal boxes at least 3.5m round internal angles. Cavity preparations were done under rubber dam with a diamond bur (100micron) with high-speed handpiece, in case of carious tissue this was removed finely. After finishing, all cavities were cleaned with air-water spray and gently air-dried in order to apply 37% phosphoric acid etchant gel on enamel and dentin. The cavities were then rinsed for 30 s with air-water spray and dried using suction to keep some moisture in dentin and a layer of bonding is applied onto the surface and light-cured. Composite material was applied in the cavities in order to create a block-out, that will eliminate undercuts and increase thickness of residual walls.

Preparations were then finished and polished with fine grain burs(60 and 40 micron respectively). After removing rubber dam, complete arch impressions were taken with a polyether material followed by disinfecting the impressions for 10 min . Provisional restorations were placed with eugenol-free temporary cement . Dental impressions and photographs are sent to dental technician for FRCFPD fabrication.

FRC FDPs were made in one dental laboratory on the full arch plaster cast. The model was first isolated with two coats of isolation medium. One unidirectional pre-impregnated E-glass fibers (Vectris- Ivoclar Vivadent, Lienchestein) was used to reinforce the veneering composite. Each bundle consists of about 4000 glass fibers, with a diameter of 1.7 mm, embedded in a PMMA/bis-GMA matrix. Before the fibers were placed on the cast, a layer of composite was applied into the interproximal-occlusal box of the abutment teeth. The fiber bundle was placed in the bed of the flowable resin using metal hand instruments.

After photo-polymerization with a halogen polymerization unit (light output: 1200 mw/cm2), the framework was veneered with a resin composite An opaque resin was used in some cases to improve the optical properties. The veneering resin composite was built incrementally; the construction was polymerized for the final time with a heat-light polymerization oven.

In the second session, after rubber dam placement and removal of provisional restorations, the teeth were cleaned with a prophylaxis brush and pumice. After try-in of the FRCFPD to check proximal contacts and marginal fit, all adhesive surfaces of the restoration were sandblasted, and then cleaned with ethanol and air-dried.

The cementation surface of the FDP was treated with resin monomer of the corresponding resin cement using a micro brush (Heliobond Ivoclar Vivadent, liechtenstein). The resin was left unpolymerized, shielded from light, for at least 5 minutes to allow the resin to penetrate and activate the IPN-phase of the polymethacrylate polymer matrix of the FRC framework.

The tooth surface was prepared for adhesion by applying a three step etch and rinse adhesive. After removal of excess resin, all restorations were cemented using a resin cement Variolink II . light-cured for 40s on each surface (lingual, labial, mesial, distal) (Astralis 10, SN 018766, Ivoclar Vivadent, light output: 1200 mW/cm2). Static and dynamic occlusion was adjusted using fine grit diamond burs. The power output of the unit was measured with a radiometer ( before the placement of each restoration. After polymerization, restoration margins were finished. Occlusion was adjusted with fine diamond burs (60- and 40-µm grit) and finally, the restoration was polished with pointed silicon polishers and abrasive polishing brushes. Patients received individual instructions to maintain plaque control.

One operator applied all the restorations who has experience in adhesive dentistry (>10 years since graduation).

ELIGIBILITY:
Inclusion criteria:

* All subjects were required to be at least 18 years old, able to read and sign the informed consent document
* Physically and psychologically able to tolerate conventional restorative procedures
* Having no active periodontal or pulpal diseases
* Having no primary caries
* Not allergic to resin-based materials
* Not pregnant or nursing
* Having antagonist teeth opposing the FRC FDP to be restored
* Willing to return for follow-up examinations as outlined by the investigators.

Exclusion Criteria:

* Patients who had more absent teeth than the tooth to be replaced in the rest of the dentition or those having diastemas were not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 1999-06; Primary Completion 2016-09 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Debonding of restoration | 15 Years
  According to USPHS criteria
Fracture of Tooth | 15 Years
  According to USPHS criteria
Fracture of Restorations | 15 Years
  According to USPHS criteria
Chipping of restoration | 15 Years
  According to USPHS criteria

SECONDARY OUTCOMES:
Secondary caries of the tooth | 15 Years
  According to USPHS criteria

IPD SHARING:
Plan to Share IPD: Undecided